CLINICAL TRIAL: NCT00012701
Title: Measuring HIV Quality of Care
Status: Completed | Type: Observational
Sponsor: US Department of Veterans Affairs (U.S. Federal Agency)
Responsible Party: Sponsor
Organization: VA Office of Research and Development (U.S. Federal Agency)
Other Study IDs: HIS 99-042
Record Dates: First submitted 2001-03-14; First posted 2001-03-16 (Estimated); Last update posted 2015-04-07 (Estimated); Status verified 2005-07

CONDITIONS: HIV Positive; Facility Level Care; Clinical Reminder
MeSH Terms: conditions — HIV Seropositivity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Group 1

SUMMARY:
The VA is the largest single provider of HIV care in the United States. The late 1990's have seen a revolution in the quality standards for this disease with the onset of Highly Active Antiretroviral Therapy (HAART) and other developments.

DETAILED DESCRIPTION:
Background:

The VA is the largest single provider of HIV care in the United States. The late 1990's have seen a revolution in the quality standards for this disease with the onset of Highly Active Antiretroviral Therapy (HAART) and other developments.

Objectives:

Our purpose in this project is to develop a method for assessing quality in two important areas of HIV care - antiretroviral medications and opportunistic infection screening and prophylaxis - and explore the determinants of high quality care in order to suggest quality improvement strategies.

Methods:

The analysis has four parts. First, it will describe the level of adherence to the indicators in VA HIV patients nationwide and compare VA HIV patients to national benchmarks. Second, it will analyze facility and patient level predictors of adherence to indicators of quality of care and compare them with the predictors in the non VA population using staged logistic regressions. Third, it will seek to validate certain indicators (e.g. HAART therapy) against clinical outcomes like hospitalization and immune status. We will also model the clinical "price" that the VA pays in suboptimal clinical outcomes as a result of current performance levels. Fourth, we will compare the performance of the facilities after one year of an intensive targeted indicator-specific feedback group versus those receiving aggregate data only.

Status:

Data analysis.

ELIGIBILITY:
Inclusion Criteria:

Facilities with HIV clinics

Exclusion Criteria:

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 1600 (Estimated)
Dates: Study Completion 2003-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Steven M. Asch, MD MPH, Principal Investigator — VA Greater Los Angeles Healthcare System, West Los Angeles, CA; Samuel A. Bozzette, MD PhD, Principal Investigator — VA San Diego Healthcare System, San Diego, CA
Locations (2):
- United States (2):
  - VA San Diego Healthcare System, San Diego, CA, San Diego, California
  - VA Greater Los Angeles Healthcare System, West Los Angeles, CA, West Los Angeles, California

REFERENCES:
- [Result] Patterson ES, Nguyen AD, Halloran JP, Asch SM. Human factors barriers to the effective use of ten HIV clinical reminders. J Am Med Inform Assoc. 2004 Jan-Feb;11(1):50-9. doi: 10.1197/jamia.M1364. Epub 2003 Oct 5. PMID 14527974
- [Result] Bozzette SA, Phillips B, Asch S, Gifford AL, Lenert L, Menke T, Ortiz E, Owens D, Deyton L. Quality Enhancement Research Initiative for human immunodeficiency virus/acquired immunodeficiency syndrome: framework and plan. HIV-QUERI Executive Committee. Med Care. 2000 Jun;38(6 Suppl 1):I60-9. doi: 10.1097/00005650-200006001-00007. PMID 10843271
- [Result] Asch SM, Fremont AM, Turner BJ, Gifford A, McCutchan JA, Mathews WM, Bozzette SA, Shapiro MF. Symptom-based framework for assessing quality of HIV care. Int J Qual Health Care. 2004 Feb;16(1):41-50. doi: 10.1093/intqhc/mzh004. PMID 15020559
- [Result] Bozzette SA, Gifford AL. The economic viability of antiretroviral adherence interventions. Am J Med. 2003 Dec 1;115(8):672-3. doi: 10.1016/j.amjmed.2003.09.023. No abstract available. PMID 14656623